CLINICAL TRIAL: NCT03016650
Title: Opioid-sparing Effect of Intravenous Ibuprofen
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muharrem Ucar (Other)
Responsible Party: Sponsor-Investigator, Muharrem Ucar, Principal Investigator, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: muharrem-1
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Analgesia; Percutaneous Nephrolithotomy
Keywords: Acetaminophen; Ibuprofen
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Active Comparator): Patients will receive 100 mL of physiologic saline with 1 g IV acetaminophen (paracetamol) 30 minutes before the end of the operation and postoperatively 6, 12 and 18 hours after percutaneous nephrolithotomy, respectively.
  Interventions: Drug: Acetaminophen
- ibuprofen (Active Comparator): Patients will receive 100 mL of physiologic saline with 800 mg IV ibuprofen 30 minutes before the end of the operation and postoperatively 6, 12 and 18 hours after percutaneous nephrolithotomy, respectively.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Patients receive 100 mL of physiologic saline with 1 g IV paracetamol 30 minutes before the end of the operation and postoperatively 6, 12 and 18 hours after PCNL
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Ibuprofen — Patients receive 100 mL of physiologic saline with 800 mg IV ibuprofen 30 minutes before the end of the operation and postoperatively 6, 12 and 18 hours after PCNL
  Other Names: Intrafen
  Arms: ibuprofen

SUMMARY:
The investigators aimed to evaluate tramadol-sparing effect of intravenous (IV) ibuprofen in patients undergoing percutaneous nephrolithotomy (PCNL).

DETAILED DESCRIPTION:
Eighty patients who will undergoing PCNL are randomized to intravenous paracetamol (n=40) and intravenous ibuprofen (n=40) groups. Patients will receive 100 mL of physiologic saline with 1 g IV paracetamol or 800 mg IV ibuprofen 30 minutes before the end of the operation and postoperatively 6, 12 and 18 hours after PCNL in the paracetamol and ibuprofen groups, respectively. Patients in both groups will receive intravenous tramadol with patient controlled analgesia device (PCA).

The visual analog scale (VAS) will used to evaluate pain intensity scores in the postoperative period.

Total tramadol consumption, mean VAS score in the 1, 8 and 24 hours, demographic variables, operative variables, and side effects will record.

ELIGIBILITY:
Inclusion Criteria:

* Study include 80 patients of American Society of Anesthesiologists (ASA) physical status I-II aged between 18-70 years who scheduled for percutaneous nephrolithotomy operation.

Exclusion Criteria:

* chronic pain,
* psychiatric disease,
* renal dysfunction,
* allergy to nonsteroidal anti-inflammatory drugs,
* history of drug addiction,
* pregnancy,
* inability to use a patient controlled analgesia (PCA) device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Morphine Consumption | postoperatively 24 hours

SECONDARY OUTCOMES:
Visual Analog Scale | postoperatively 30 minute, 2, 4, 6,12 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Muharrem Ucar, Principal Investigator — İnonu University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maghsoudi R, Tabatabai M, Radfar MH, Movasagi G, Etemadian M, Shati M, Amjadi M. Opioid-sparing effect of intravenous paracetamol after percutaneous nephrolithotomy: a double-blind randomized controlled trial. J Endourol. 2014 Jan;28(1):23-7. doi: 10.1089/end.2013.0267. Epub 2013 Oct 17. PMID 23952097